CLINICAL TRIAL: NCT00916474
Title: EXTEND: A 3-Year, Virology Follow up Study in Subjects Previously Treated With Telaprevir in Select Clinical Studies
Brief Title: Virology Follow up Study in Subjects Previously Treated With Telaprevir
Status: Completed | Type: Observational
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: VX08-950-112
Record Dates: First submitted 2009-06-04; First posted 2009-06-09 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort A: Observational follow-up study to assess long-term response to telaprevir and to evaluate changes in Hepatitis C virus over time
  Interventions: Drug: telaprevir
- Cohort B: Observational follow-up study to assess long-term response to telaprevir and to evaluate changes in Hepatitis C virus over time
  Interventions: Drug: telaprevir

INTERVENTIONS:
Drug: telaprevir

SUMMARY:
Observational follow-up study to assess long-term response to telaprevir and to evaluate changes in Hepatitis C virus over time.

ELIGIBILITY:
Inclusion Criteria:

* Received at least 1 dose of telaprevir-based treatment in 1 of the following clinical studies: VX05-950-104, VX05-950-104EU, VX06-950-106, VX06-950-107, VX07-950-108, VX08-950-111, or VX-950-TiDP24-C216
* Have baseline HCV viral sequencing data available from previous telaprevir study

Exclusion Criteria:

* May not be currently participating in the antiviral follow-up period of an ongoing telaprevir trial. (Note: Subjects who have completed the required antiviral follow-up period but are still participating in the collection of patient-reported outcomes data for their previous telaprevir study may be eligible.)
* For subjects participating in ongoing studies at the time of enrollment, have more than 90 elapsed days between the database lock or unblinding in the previous telaprevir study and Day 1 in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have previously received at least 1 dose of telaprevir-based treatment (telaprevir plus peginterferon alfa 2a [Peg IFN-alfa-2a] with or without ribavirin [RBV]) in 1 of the following clinical studies: VX05-950-104, VX05 950-104EU, VX06-950-106, VX06-950-107, VX07-950-108, VX08-950-111, and VX-950-TiDP24-C216.
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2009-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who maintain undetectable HCV RNA over time after achieving an SVR following telaprevir-based treatment | 3 years
Change in HCV variants with decreased sensitivity to telaprevir over time in subjects failing to achieve an SVR following telaprevir-based treatment | 3 years

SECONDARY OUTCOMES:
Change in HCV variants with decreased sensitivity to telaprevir over time in subjects with late relapse | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (41):
- United States (25):
  - Alabama, Birmingham, Alabama
  - California, Coronado, California
  - California, Los Angeles, California
  - California, San Francisco, California
  - Colorado, Denver, Colorado
  - Colorado, Englewood, Colorado
  - Florida, Gainsville, Florida
  - Florida, Jacksonville, Florida
  - Florida, Miami, Florida
  - Georgia, Altanta, Georgia
  - Maryland, Baltimore, Maryland
  - Massachusetts, Boston, Massachusetts
  - Michigan, Novi, Michigan
  - Missouri, St Louis, Missouri
  - New Mexico, Albuquerque, New Mexico
  - New York, Manhasset, New York
  - New York, New York, New York
  - North Carolina, Chapel Hill, North Carolina
  - North Carolina, Durham, North Carolina
  - Ohio, Cincinnati, Ohio
  - South Carolina, Columbia, South Carolina
  - Texas, Houston, Texas
  - Texas, San Antonio, Texas
  - Virginia, Fairfax, Virginia
  - Virginia, Falls Church, Virginia
- Canada (2):
  - Canada, Vancouver, British Columbia
  - Canada, Toronto, Ontario
- France (5):
  - France, Clichy
  - France, Marseille
  - France, Paris
  - France, Pessac
  - France, Vandœuvre-lès-Nancy
- Germany (8):
  - Germany, Berlin
  - Germany, Cologne
  - Germany, Frankfurt
  - Germany, Freiburg im Breisgau
  - Germany, Hamburg
  - Germany, Hanover
  - Germany, Munich
  - Germany, Wien
- Puerto Rico, Santurce, Puerto Rico